CLINICAL TRIAL: NCT07095127
Title: An Open-label, Intra-participant Dose Escalation Study to Evaluate the Safety, Tolerability, and Efficacy of Intravenous NVG-2089 in Participants With Immune Thrombocytopenia
Brief Title: Safety, Tolerability, and Efficacy of NVG-2089 in Participants With Immune Thrombocytopenia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nuvig Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NVG-2089-200
Record Dates: First submitted 2025-07-11; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Immune Thrombocytopenia (ITP)
Keywords: Immune Thrombocytopenia, ITP
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- NVG-2089 (Experimental): NVG-2089
  Interventions: Drug: NVG-2089

INTERVENTIONS:
Drug: NVG-2089 — Study Treatment

SUMMARY:
The purpose of the study is to evaluate the safety of NVG-2089 and to evaluate how well patients respond to this investigational treatment. NVG-2089 is a new drug that is being developed for treating patients with ITP. NVG-2089 is designed to mimic the effects of a protein called IVIg. NVG-2089 is designed to help the immune system by attaching (binding) to certain receptors in the body and activating them, which helps reduce inflammation and supports how the immune system works.

ELIGIBILITY:
Inclusion Criteria:

* Males and female participants, age 18 to 80 years at time of screening.
* Diagnosis of persistent (>3 months and ≤12 months), or chronic (>12 months) primary ITP. If the participant has received prior treatment for ITP, they must have a history of response to at least one previous therapy (defined as increase in platelet count to ≥ 50,000 cells/mm3 with an increase of ≥ 20,000 cells/mm3 relative to platelet count prior to treatment).
* Asymptomatic or with minor mucocutaneous bleeding AND platelet count of ≥ 20,000 to ≤50,000 cells/mm3, measured on 2 occasions. At least one measurement should be obtained during screening. Documented historical platelet count obtained within 4 weeks prior to screening will also be acceptable for one of the two readings.
* (For US only) If at least one screening platelet count >30,000 cells/ mm3 and <50,000 cells/mm3, the participant must be on at least 1 other treatment for ITP with insufficient response as evidenced by platelet count <50,000 cells/ mm3.
* If participant has received prior IVIg therapy participant must have shown a sufficient platelet response (doubling from baseline platelet count within 7 days of IVIg infusion) and must not have lost response to IVIg therapy while on treatment.
* Female participants of childbearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day 1.
* Female participants who are sexually active with a male partner of reproductive potential must use double contraception (including a barrier contraceptive and another method) from at least 28 days prior to Screening and for 90 days after last dose of study drug; female participants must also refrain from oocyte donation for the purpose of reproduction during this period. Exceptions are made for surgically sterile participants, or post-menopausal females (defined as 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum follicle -stimulating hormone levels >40 mIU/mL or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy). Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the participant.
* Male participants with female partners who are of reproductive potential must agree to the use of highly effective, barrier contraception for the duration of the study, and for 90 days after the last dose of study drug.
* Participant is capable or has a legally authorized representative(s) (LAR[s]) capable of providing a signed informed consent which includes compliance with the requirements and restrictions listed in the ICF.

Exclusion Criteria:

* Secondary forms of ITP (e.g., ITP secondary to infection, autoimmune diseases, lymphoproliferative diseases and medications).
* History of splenectomy.
* History of malignancy, unless the participant received treatment with curative intent. Participants with fully excised non-melanoma skin cancer or cervical cancer are allowed.
* History of solid organ transplant.
* Planned or anticipated medical or surgical procedure, including dental procedure, during the timeframe of the study conduct.
* Clinically significant active or chronic uncontrolled bacterial, viral, or fungal infection at screening, including active viral infection at screening.
* Any medical condition that, in the opinion of the investigator, would interfere with study evaluations or procedures, and/or put the participant at increased risk.
* ECG findings of QTcF > 450 msec (males) or > 470 msec (females), poorly controlled atrial fibrillation or other clinically significant abnormalities.
* Other significant organ dysfunction, including but not limited to, hematologic, renal, or hepatic dysfunction, as evidenced by:

  1. Absolute neutrophil count ≤ 1.5 x 109 /L
  2. Hemoglobin (Hgb) < 9 g/dL
  3. Aspartate aminotransaminase (AST) and/or alanine aminotransferase (ALT) ≥ 2 x the upper limit of normal (ULN),
  4. Albumin ≤ 3 g/dL
  5. Total bilirubin ≥ 1.5 x ULN
  6. Estimated glomerular filtration rate < 50 mL/min/1.73m2 using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) method
* Any of the following at screening:

  1. Active Hepatitis B Virus (HBV): Hepatitis surface antigen (HBsAg) positive
  2. Active Hepatitis C Virus (HCV): serology positive for HCV-antibody
  3. Human Immunodeficiency Virus (HIV) positive serology
* Transfusion of blood, blood products (including immune globulin), or plasmapheresis within 4 weeks prior to screening.
* Change in current ITP therapy (e.g., prednisone, methylprednisone, mycophenolate, dapsone, danazol, azathioprine, or TPO receptor agonist) or dose within 4 weeks prior to screening.
* Receipt of dexamethasone within 4 weeks prior to screening.
* Receipt of rituximab or an anti-CD20 agent within 6 months prior to screening.
* Receipt of an neonatal Fc receptor (FcRn) inhibitor within 12 weeks prior to screening.
* Receipt of IVIg within 4 weeks prior to screening.
* Receipt of another investigational drug within 4-weeks or 5 half-lives (whichever is longer) prior to screening.
* Concurrent treatment with other monoclonal antibody and/or Fc therapies.
* Current or past history (within 12 months of screening) of alcohol, drug, or medication abuse. Positive urine drug screen at screening visit.
* Pregnant or lactating women and those intending to become pregnant during the study or are unwilling to apply an effective birth control method (such as implants, injectables, combined oral contraceptives, intrauterine devices [IUDs], sexual abstinence, or vasectomized partner) up to 90 days after last study drug administration.
* Poor venous access.
* A known allergy to study drug and/or any of its components.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate incidence, nature and severity of Treatment Emergent Adverse Events (TEAEs) | From enrollment to end of treatment Day 85
Evaluate incidence, nature and severity of Serious Adverse Events (SAEs) | From enrollment to end of treatment Day 85

SECONDARY OUTCOMES:
Percent of participants achieving a response. | From enrollment to Treatment Day 57-64
  * For participants with a baseline platelet count between 20,000 to 30,000 cells/mm3 a response is defined as a doubling of the baseline platelet count or a platelet count of ≥50,000 cells/mm3;
  * For participants with a baseline platelet count between 30,000 to 50,000 cell/mm3, a response is defined as doubling of platelet count from baseline or a platelet count of ≥80,000 cells/mm3
  * Increase in platelet count of ≥20,000 cells/mm3 from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Nuvig Site, Westbury, New York, United States

IPD SHARING:
Plan to Share IPD: No